CLINICAL TRIAL: NCT06137209
Title: Assessment of Colonisation and Skin Quality Parameter Improvement by Probiotic Micrococcus Luteus Q24 Serum in Healthy Adults
Brief Title: Colonization of Skin by M. Luteus Q24 Probiotic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BLIS Technologies Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BLTCT2022/10
Record Dates: First submitted 2023-11-05; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Microbial Colonization
Keywords: probiotics
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups applying serum containing Micrococcus luteus Q24 at a low or higher dose of probiotic.
  Group A: Probiotic Micrococcus luteus Q24 serum (dose:1e7 colony forming units per application of serum).
  Group B: Probiotic Micrococcus luteus Q24 serum (dose:1e6 colony forming units per application of serum)
Who Masked: Participant, Investigator
Masking Description: A Staff member will be assigned to distribute blinded samples. The investigator will not be aware of the dose groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group A: Blis Q24 Serum at 1e7 cfu/ dose (Active) (Active Comparator): Group A: Probiotic Micrococcus luteus Q24 serum (dose: 1e7 colony forming units per application)
  Interventions: Other: Active Comparator: Study Group A: Blis Q24 Serum at higher dose
- Study Group B: Blis Q24 Serum at 1e6 cfu/ dose (Active) (Active Comparator): Group B: Probiotic Micrococcus luteus Q24 serum (dose: 1e6 colony forming units per application)
  Interventions: Other: Active Comparator: Study Group B: Blis Q24 Serum at lower dose

INTERVENTIONS:
Other: Active Comparator: Study Group A: Blis Q24 Serum at higher dose — Active Comparator: Study Group A: Blis Q24 Serum at 1e7 cfu/ dose (Active)
  Arms: Study Group A: Blis Q24 Serum at 1e7 cfu/ dose (Active)
Other: Active Comparator: Study Group B: Blis Q24 Serum at lower dose — Active Comparator: Study Group B: Blis Q24 Serum at 1e6 cfu/ dose (Active)
  Arms: Study Group B: Blis Q24 Serum at 1e6 cfu/ dose (Active)

SUMMARY:
The purpose of this study is to evaluate the skin quality improvement and colonization efficacy following the application of probiotic Micrococcus luteus Q24 (BLIS Q24) to the face from a serum format in healthy adults.

DETAILED DESCRIPTION:
This is a randomized double-blind baseline controlled pilot study with no crossover for the assessment of any changes to the microbial make-up of the skin (The local skin microbiome), detection of colonization by the probiotic bacterium (BLIS Q24) on the skin and to evaluate the changes in skin quality parameters following topical application of probiotic in a serum format.

ELIGIBILITY:
Inclusion criteria:

1. In general good health 18 - 80 years of age.
2. Practice good general body hygiene.

Exclusion criteria:

1. Have a history of autoimmune disease or are immunocompromised (have a weakened immune system).
2. Are on concurrent antibiotic therapy or regular antibiotic use within the last 1 week.
3. People with allergies or sensitivity to dairy.
4. People with an open wound on the Blis Q24 application sites.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2023-11-22 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in microbial composition following application of 1e7 cfu per dose Micrococcus luteus Q24 in serum from Day 0 (baseline) to 11 days | Time Frame: 11 days post intervention
  Study will determine the change in microbial composition following the application of 1e7 cfu per dose serum containing Micrococcus luteus Q24 serum at one body site (face). The statistical analysis will be carried out to compare the participants skin swab data from baseline to 11 days across one site with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software. Analysis will be performed using bacterial genome sequence analysis of the skin swab samples collected.
Change in skin quality parameters following application of 1e7 cfu per dose Micrococcus luteus Q24 in serum from Day 0 (baseline) to 11 days | Time Frame: 11 days post intervention
  Study will determine the change in skin quality parameters following the application of 1e7 cfu per dose serum containing Micrococcus luteus Q24 serum at one body site (face). The statistical analysis will be carried out to compare the participants skin quality data from baseline to 11 days across one site with a level of significance of p<0.05. Overall skin quality data based on percentage of population will also be analyzed using appropriate statistical analysis software. Analysis will be performed using a portable handheld skin analyzer device that measures key cosmetic parameters such as hydration, pores, spots and wrinkles.
Change in microbial composition following application of 1e6 cfu per dose Micrococcus luteus Q24 in serum from Day 0 (baseline) to 11 days | Time Frame: 11 days post intervention
  Study will determine the change in microbial composition following the application of 1e6 cfu per dose serum containing Micrococcus luteus Q24 serum at one body site (face). The statistical analysis will be carried out to compare the participants skin swab data from baseline to 11 days across one site with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software. Analysis will be performed using bacterial genome sequence analysis of the skin swab samples collected.
Change in skin quality parameters following application of 1e6 cfu per dose Micrococcus luteus Q24 in serum from Day 0 (baseline) to 11 days | Time Frame: 11 days post intervention
  Study will determine the change in skin quality parameters following the application of 1e6 cfu per dose serum containing Micrococcus luteus Q24 serum at one body site (face). The statistical analysis will be carried out to compare the participants skin quality data from baseline to 11 days across one site with a level of significance of p<0.05. Overall skin quality data based on percentage of population will also be analyzed using appropriate statistical analysis software. Analysis will be performed using a portable handheld skin analyzer device that measures key cosmetic parameters such as hydration, pores, spots and wrinkles.
Change in microbial composition following application of 1e7 cfu per dose Micrococcus luteus Q24 in serum from Day 0 (baseline) to 30 days | Time Frame: 30 days post intervention
  Study will determine the change in microbial composition following the application of a serum containing 1e7 cfu per dose of Micrococcus luteus Q24 serum at one body site (face). The statistical analysis will be carried out to compare the participants skin swab data from baseline to 30 days across one site with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software. Analysis will be performed using bacterial genome sequence analysis of the skin swab samples collected.
Change in skin quality parameters following application of 1e7 cfu per dose Micrococcus luteus Q24 in serum from Day 0 (baseline) to 30 days | Time Frame: 30 days post intervention
  Study will determine the change in skin quality parameters following the application of 1e7 cfu per dose serum containing Micrococcus luteus Q24 serum at one body site (face). The statistical analysis will be carried out to compare the participants skin quality data from baseline to 30 days across one site with a level of significance of p<0.05. Overall skin quality data based on percentage of population will also be analyzed using appropriate statistical analysis software. Analysis will be performed using a portable handheld skin analyzer device that measures key cosmetic parameters such as hydration, pores, spots and wrinkles.
Change in microbial composition following application of 1e6 cfu per dose Micrococcus luteus Q24 in serum from Day 0 (baseline) to 30 days | Time Frame: 30 days post intervention
  Study will determine the change in microbial composition following the application of a serum containing 1e6 cfu per dose of Micrococcus luteus Q24 serum at one body site (face). The statistical analysis will be carried out to compare the participants skin swab data from baseline to 30 days across one site with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software. Analysis will be performed using bacterial genome sequence analysis of the skin swab samples collected.
Change in skin quality parameters following application of 1e6 cfu per dose Micrococcus luteus Q24 in serum from Day 0 (baseline) to 30 days | Time Frame: 30 days post intervention
  Study will determine the change in skin quality parameters following the application of 1e6 cfu per dose serum containing Micrococcus luteus Q24 serum at one body site (face). The statistical analysis will be carried out to compare the participants skin quality data from baseline to 30 days across one site with a level of significance of p<0.05. Overall skin quality data based on percentage of population will also be analyzed using appropriate statistical analysis software. Analysis will be performed using a portable handheld skin analyzer device that measures key cosmetic parameters such as hydration, pores, spots and wrinkles.
Change in microbial composition post 7 days of last application of 1e7 cfu of Micrococcus luteus Q24 in serum. | Time Frame: 7 days post last intervention
  Study will determine the change in microbial composition following the application of a serum containing 1e7 cfu per dose of Micrococcus luteus Q24 serum at one body site (face). The statistical analysis will be carried out to compare the participants skin swab data at Day 37 (i.e. post 7 days from last application) across one site with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software. Analysis will be performed using bacterial genome sequence analysis of the skin swab samples collected.
Change in skin quality parameters post 7 days of last application of 1e7 cfu of Micrococcus luteus Q24 in serum. | Time Frame: 7 days post last intervention
  Study will determine the change in skin quality parameters following the application of a serum containing 1e7 cfu per dose of Micrococcus luteus Q24 serum at one body site (face). The statistical analysis will be carried out to compare the participants skin swab data at Day 37 (i.e. post 7 days from last application) across one site with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software. Analysis will be performed using a portable handheld skin analyzer device that measures key cosmetic parameters such as hydration, pores, spots and wrinkles.
Change in microbial composition post 7 days of last application of 1e6 cfu of Micrococcus luteus Q24 in serum. | Time Frame: 7 days post last intervention
  Study will determine the change in microbial composition following the application of a serum containing 1e6 cfu per dose of Micrococcus luteus Q24 serum at one body site (face). The statistical analysis will be carried out to compare the participants skin swab data at Day 37 (i.e. post 7 days from last application) across one site with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software. Analysis will be performed using bacterial genome sequence analysis of the skin swab samples collected.
Change in skin quality parameters post 7 days of last application of 1e6 cfu of Micrococcus luteus Q24 in serum. | Time Frame: 7 days post last intervention
  Study will determine the change in skin quality parameters following the application of a serum containing 1e6 cfu per dose of Micrococcus luteus Q24 serum at one body site (face). The statistical analysis will be carried out to compare the participants skin swab data at Day 37 (i.e. post 7 days from last application) across one site with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software. Analysis will be performed using a portable handheld skin analyzer device that measures key cosmetic parameters such as hydration, pores, spots and wrinkles.

CONTACTS AND LOCATIONS:
Locations (1):
- Blis Technologies Ltd, Dunedin, Otago, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Data and information in the protocol and the clinical study report will be shared to other researchers and/or in publications in due course.
Supporting Information: Study Protocol, CSR
Time Frame: Study report 3 months after completion of the study.
Access Criteria: Summary study report will be shared by the Principal Investigator upon request if not published in public literature.

REFERENCES:
- [Background] van Rensburg JJ, Lin H, Gao X, Toh E, Fortney KR, Ellinger S, Zwickl B, Janowicz DM, Katz BP, Nelson DE, Dong Q, Spinola SM. The Human Skin Microbiome Associates with the Outcome of and Is Influenced by Bacterial Infection. mBio. 2015 Sep 15;6(5):e01315-15. doi: 10.1128/mBio.01315-15. PMID 26374122
- [Background] Bourdichon F, Casaregola S, Farrokh C, Frisvad JC, Gerds ML, Hammes WP, Harnett J, Huys G, Laulund S, Ouwehand A, Powell IB, Prajapati JB, Seto Y, Ter Schure E, Van Boven A, Vankerckhoven V, Zgoda A, Tuijtelaars S, Hansen EB. Food fermentations: microorganisms with technological beneficial use. Int J Food Microbiol. 2012 Mar 15;154(3):87-97. doi: 10.1016/j.ijfoodmicro.2011.12.030. Epub 2011 Dec 31. PMID 22257932